CLINICAL TRIAL: NCT04624542
Title: Relation Between Femoral Nerve Conduction Velocity and Its Mechanosensitivity Changes Among Individual With Patellofemoral Pain Syndrome
Brief Title: Relation Between Femoral Nerve Conduction Velocity and Its Mechanosensitivity Changes Among Patellofemoral Pain Syndrome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nabil Abdo Abdellah Mohamed, lecturer of orthopedic physiotherapy /faculty of physical therapy cairo university, Cairo University
Other Study IDs: NCV for PFPS
Record Dates: First submitted 2020-11-05; First posted 2020-11-12 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Patello Femoral Syndrome
Keywords: femoral nerve conduction velocity
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group 1: Thirty individuals diagnosed with unilateral chronic PFPS from both genders and age between 18-35 years who will be referred from an orthopedic surgeon.
  Interventions: Device: Electromyographic device
- control group: -30 healthy active individuals ranging from 18-36 yrs as a controlled group
  Interventions: Device: Electromyographic device

INTERVENTIONS:
Device: Electromyographic device — the EMG machine will be used to measure NCV of femoral nerve within individuals with PFPS

SUMMARY:
1. to investigate the relation between NCV of femoral nerve and other dependent variables such as ( pain & limited hip extension ROM )in patients with PFPS .
2. to predict using the NCV as a method for assessment femoral nerve mechanosensitivity in those with PFPS

DETAILED DESCRIPTION:
Patellofemoral pain syndrome (PFPS) is considered one of the most common condition affecting young active populations, it accounts for about 40% of individuals complaining from knee pain.PFPS is the anterior or retro patellar pain that can be precipitated by some daily activities such as ascending and descending stairs, kneeling, squatting or performing everyday tasks. Individuals with PFPS can experience a history of cracking or popping sounds when changing position or climbing stairs and also experience pain during repeated knee flexion. In a previous study conducted by Jensen et al .(2008),they observed that individuals with PFPS experienced symptoms that are related to neural compromise like patellar numbness and reduced ability to differentiate between different thermal stimulus .so PFPS may be related to neurological impairments or dysfunction.

Femoral slump test can be used in examining the neurodynamic responses in individuals with anterior knee pain which has a specificity of more than 75% in testing neural mechanosensitivity In a study conducted by Lin et al (2014) that examine the hip extension range of motion (ROM) and mechanical sensitivity of femoral nerve as a neurodynamic response in individuals with PFPS , they proposed that 30% of them have decrease hip extension ROM and increased mechanosensitivity comparison with healthy individuals. The current management of the patellofemoral pain support using open- and closed-chain exercises, strengthening, stretching, aerobic exercise, patellofemoral and tibiofemoral mobilizations, patellar taping, highintensity NMES, neuromuscular training, and gait retraining as a multi modal treatment for PFPS. Despite these methods result in significant improvement, other few patients reported some residual symptoms Hung et al .,(2015) have encouraged that using the femoral nerve mobilization as a neurodynamic management for treating PFPS patients especially those with postive femoral slump test , and testing the hip extension range of motion as a reference of improvement previous studies reported the presence of neurogenic dysfunction model to PFPS but most of these scientific researches lack the presence of the gold standard and objective method for identifying the neurogenic patellofemoral pain

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria screened by the clinicians was pain during patellar palpation. In addition, subjects needed to fulfill all of the following requirements to be included in the PFP group:

  1. Patient reporting symptoms of insidious onset and duration of at least 1 month (de Oliveira et al .,2016)
  2. Peri- or retropatellar pain during at least 2 of the following activities: squatting, prolonged sitting, kneeling, running, jumping and climbing stairs (Vegstein et al., 2019)
  3. Worst pain level in the previous month of up to 3cm on a 10cm numerical rating scale (NRS). (de Oliveira et al .,2016)
  4. BMI 25-30 kg/cm2 (Nouri F et al .,2019)
  5. Showing 2 or more positive signs on the following clinical tests:

Clarke's sign, Waldron test, active patellar grind test, patellar compression test ,and palpation of the medial/lateral articular border of the patella.(hung et al., 2015) To be included in the control group CG, participants could not present any signs or symptoms of PFP or other musculoskeletal conditions

Exclusion Criteria:

* 1) inflammatory process of lower limb (Lin et al., 2014 ) 2) patellar tendon or meniscus tears (hung et al., 2015) 3) bursitis and ligament tears (hung et al., 2015) 4) Those who had undergone knee surgery, oral steroids and knee injection were excluded from this study (Vegstein et al., 2019) 5) lower back dysfunction such as disc lesion , sciatica or spondylolisthesis (Lin et al., 2014 ) 6) participants that had undergone physiotherapy during the preceding 6 months (de Oliveira et al .,2016)

Ages: 18 Years to 36 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants recruitment to this study will be conducted over 2 steps process. In the first step, all participants in the experimental group that will be referred from an orthopedic surgeon with diagnosis of unilateral PFPS to the outpatient clinic at Cairo University hospital at kasr el ainy
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
the patellofemoral pain | 6 months
  pain will be measured by using the Pain numeric rating scale (NRS)

SECONDARY OUTCOMES:
range of hip extension | 6 month
  ROM will be measured using universal goniometer

CONTACTS AND LOCATIONS:
Overall Officials: nabil ab abdo, Study Director — PHD faculty of physical therapy Cairo university

IPD SHARING:
Plan to Share IPD: Undecided
the data include his /her name ,age, sex , demographic data including (height,weight &BMI ) and the phone number and address with ID number

REFERENCES:
- [Background] Fredericson M, Yoon K. Physical examination and patellofemoral pain syndrome. Am J Phys Med Rehabil. 2006 Mar;85(3):234-43. doi: 10.1097/01.phm.0000200390.67408.f0. PMID 16505640
- [Background] Fredericson M, Powers CM. Practical management of patellofemoral pain. Clin J Sport Med. 2002 Jan;12(1):36-8. doi: 10.1097/00042752-200201000-00010. No abstract available. PMID 11854587
- [Background] Jensen R, Kvale A, Baerheim A. Is pain in patellofemoral pain syndrome neuropathic? Clin J Pain. 2008 Jun;24(5):384-94. doi: 10.1097/AJP.0b013e3181658170. PMID 18496302
- [Background] Jensen R, Hystad T, Kvale A, Baerheim A. Quantitative sensory testing of patients with long lasting Patellofemoral pain syndrome. Eur J Pain. 2007 Aug;11(6):665-76. doi: 10.1016/j.ejpain.2006.10.007. Epub 2007 Jan 3. PMID 17204440
- [Background] Eliav E, Benoliel R, Tal M. Inflammation with no axonal damage of the rat saphenous nerve trunk induces ectopic discharge and mechanosensitivity in myelinated axons. Neurosci Lett. 2001 Sep 21;311(1):49-52. doi: 10.1016/s0304-3940(01)02143-7. PMID 11585565
- [Background] Sanchis-Alfonso V, Rosello-Sastre E. Immunohistochemical analysis for neural markers of the lateral retinaculum in patients with isolated symptomatic patellofemoral malalignment. A neuroanatomic basis for anterior knee pain in the active young patient. Am J Sports Med. 2000 Sep-Oct;28(5):725-31. doi: 10.1177/03635465000280051801. PMID 11032232
- [Background] Heintjes E, Berger MY, Bierma-Zeinstra SM, Bernsen RM, Verhaar JA, Koes BW. Exercise therapy for patellofemoral pain syndrome. Cochrane Database Syst Rev. 2003;(4):CD003472. doi: 10.1002/14651858.CD003472. PMID 14583980
- [Result] Smith BE, Selfe J, Thacker D, Hendrick P, Bateman M, Moffatt F, Rathleff MS, Smith TO, Logan P. Incidence and prevalence of patellofemoral pain: A systematic review and meta-analysis. PLoS One. 2018 Jan 11;13(1):e0190892. doi: 10.1371/journal.pone.0190892. eCollection 2018. PMID 29324820